CLINICAL TRIAL: NCT06224699
Title: Clinical and Antimicrobial Effectiveness of a Toothpaste With Sodium Carbonate in Patients With Gingivitis
Brief Title: Toothpaste With Sodium Carbonate in Patients With Gingivitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Gaetano Isola, Associate Professor, University of Catania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 149/22/PO
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Gingivitis; Periodontal Diseases
MeSH Terms: conditions — Gingivitis; Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: The study was designed as a double-blind randomized controlled trial (RCT) with 2 parallel groups of individuals with gingivitis
Who Masked: Participant, Investigator
Masking Description: Sealed envelopes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Use of toothpaste with sodium carbonate 67%
  Interventions: Drug: Toothpaste Product
- Control (Placebo Comparator): Use of toothpaste without sodium carbonate 67%
  Interventions: Drug: Toothpaste Product

INTERVENTIONS:
Drug: Toothpaste Product — Use of toothpaste with or without sodium carbonate at 67%

SUMMARY:
Sodium carbonate has several properties that may be beneficial in the management of bacterial biofilm in gingivitis patients. The aim of this RCT study is to clinically evaluate the clinical properties of two toothpaste containing Sodium carbonate 67% and fluoride toothpaste that contains no bicarbonate on patients with gengivitis.

DETAILED DESCRIPTION:
Sodium carbonate has several properties that may be beneficial in the management of bacterial biofilm in both gingivitis and periodontitis patients. The aim of this RCT study is to clinically evaluate the clinical properties of two toothpaste containing sodium carbonate at 67% or no sodium carbonate at 67% at 6-month follow-up in patients with gingivits. The study was designed as a double-blind randomized controlled trial (RCT) with 2 parallel groups of individuals.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with gingivitis according to the EFP/AAP 2017 criteria.

Exclusion Criteria:

* Periodontal treatment, antibiotics, NSAIDs, immunosuppressants during the last 6 months.
* Pregnancy.
* Systemic diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Gingival index (1-4) | 6-months
  Gingival index reduction

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Policlinico Catania, Catania, Italy

IPD SHARING:
Plan to Share IPD: Yes
Study results
Supporting Information: Study Protocol
Time Frame: 1-year
Access Criteria: Pubmed